CLINICAL TRIAL: NCT00993681
Title: A Phase Three, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy of the Travelers' Diarrhea Vaccine System
Brief Title: Travelers' Diarrhea (TD) Vaccine Pivotal Efficacy Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intercell USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ELT301; EudraCT Number: 2008-008726-75
Record Dates: First submitted 2009-10-08; First posted 2009-10-12 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Travelers' Diarrhea
Keywords: Prevention of Travelers' Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 900 subjects will receive a two vaccination regimen with an LT patch
  Interventions: Biological: TD Vaccine System
- 2 (Placebo Comparator): 900 subjects will receive a two vaccination regimen with a placebo patch
  Interventions: Biological: TD Vaccine System

INTERVENTIONS:
Biological: TD Vaccine System — heat labile enterotoxin of E. coli (LT)
  Arms: 1
Biological: TD Vaccine System — placebo
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy of the Travelers' Diarrhea Vaccine System to actively immunize against Enterotoxigenic Escherichia coli disease in a field setting.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years of age at date of first vaccination
* Good health as determined by medical history and physical inspection
* Females of child-bearing potential must have a negative pregnancy test prior to first vaccination in teh Country of Origin; females of child-bearing potential must agree not to become pregnant throughout the duration of the study
* Subjects must have planned travel to an area within 3 hours traveling distance of Mexico City, Cuernavaca, Guadalajara, Oaxaca, or San Miguel de Allende, Mexico or Antigua, Quezaltenango, Guatemala City, or Solola, Guatemala for a minimum duration of stay 7 days (no maximum stay is specified for inclusion).
* Subject must be able to communicate in English

Exclusion Criteria:

* Abnormalities as determined by the Investigator/clinician during physical inspection
* Participated in research involving investigational product within 30 days before planned date of first vaccination
* Ever received LT, ETEC, or cholera vaccine
* History of diarrhea while traveling to a developing country within the last year
* Women who are pregnant or breastfeeding
* Clinically significant underlying enteric, pulmonary, cardiac, liver or renal disease
* History of Irritable Bowel Syndrome
* Seizure disorder within the last year
* Current use of immunosuppressive therapy (excluding inhaled steroids) or current immunodeficiency
* Known or suspected alcohol abuse or illicit drug use within the last year
* Medical history of HIV, HBV, or HCV
* An employee of a study site
* Known allergies to any component of the vaccine, including adhesives
* Planned use of antibiotics with known activity against gram negative facultative anaerobes
* Planned use of antacids, antidiarrheals, loperamide, bismuth subsalicylate, diphenoxylate or similar during the surveillance phase of the study
* An employee of Intercell (global) or an immediate family member

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2036 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Incidence of cases with vaccine preventable outcome | Day 17 (17 days after arrival in destination country)

SECONDARY OUTCOMES:
The incidence of moderate/severe diarrhea | Day 17 (17 days after arrival in destination country)
Total unformed stool frequency from diarrheal episodes | Day 17 (17 days after arrival in destination country)
Total duration of diarrheal episodes | Day 17 (17 days after arrival in destination country)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert L Dupont, MD, Principal Investigator — Center for Infectious Diseases, The University of Texas Health Sciences Center at Houston
Locations (20):
- Germany (4):
  - University Medical Centre Hamburg-Eppendorf, Hamburg, Hamburg
  - Ludwig-Maximilians-Universitat Abt. for Infektions and Tropenmedizin, München, Munchen
  - Klinik for Gastroenterologie & Infektiologie, Potsdam, Potsdam
  - Berliner Centrum Reise & Tropenmedizin, Berlin, State of Berlin
- Guatemala (4):
  - Trek Study Antigua, Antigua, Departamento de Guatemala
  - Isthmian Medical Research Guatemala S.A., Guatemala City, Departamento de Guatemala
  - SAMI-SSAPFORFAM Consultorio Privado, Sololá, Departamento de Sololá
  - Consultorio Privado, Quetzaltenango, Quezaltenango CP
- Mexico (5):
  - Roberto Maxwell's Office, San Miguel de Allende, Guanajuato
  - Consultorio Privado Torre Medica San Javier, Guadalajara, Jalisco
  - Mexican Institute of Clinical Research (IMIC), Mexico City, Mexico City
  - Internal Medicine Trek Study Cuernavaca, Cuernavaca, Morelos
  - Hospital Reforma, Oaxaca City, Oaxaca
- United Kingdom (7):
  - Synexus Thames Valley Clinical Research Center, Reading, Berkshire
  - Synexus Midlands Clinical Research Center, Edgbaston, Birmingham
  - Synexus Lancashire Clinical Research Center, Chorley, Lancashire
  - Hospital for Tropical Diseases, London, London
  - Guy's Drug Research Unit, London Bridge, London
  - Bio-Kinetic Europe Ltd, Belfast, Northern Ireland
  - Synexus Scotland Clinical Research Center, Glasgow, Scottland

REFERENCES:
- [Derived] Behrens RH, Cramer JP, Jelinek T, Shaw H, von Sonnenburg F, Wilbraham D, Weinke T, Bell DJ, Asturias E, Pauwells HL, Maxwell R, Paredes-Paredes M, Glenn GM, Dewasthaly S, Stablein DM, Jiang ZD, DuPont HL. Efficacy and safety of a patch vaccine containing heat-labile toxin from Escherichia coli against travellers' diarrhoea: a phase 3, randomised, double-blind, placebo-controlled field trial in travellers from Europe to Mexico and Guatemala. Lancet Infect Dis. 2014 Mar;14(3):197-204. doi: 10.1016/S1473-3099(13)70297-4. Epub 2013 Nov 29. PMID 24291168